CLINICAL TRIAL: NCT04372420
Title: Recombinant Human Bone Morphogenetic Protein-2 In Absorbable Sponge Vs Platelet Rich Fibrin (PRF) In Grade Ii Furcation Defects - A Randomized Controlled Trial
Brief Title: Bone Morphogenetic Protein-2 In Grade II Furcation Defects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Principal Investigator, SVS Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVSIDS/PERIO/3/2017
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2019-12

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Group A- RhBMP-2 absorbable sponge is placed in grade II furcation and Group B- PRF is placed in the grade II furcation
Who Masked: Participant, Outcomes Assessor
Masking Description: participant and outcome assessor are masked from the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RhBMP-2 (Active Comparator): RhBMP-2 belongs to TGF-β super family with osteoinductive property which is capable of promoting bone formation
  Interventions: Drug: RhBMP-2 absorbable sponge in grade II furcation
- PLATELET RICH FIBRIN (Placebo Comparator): Platelet rich fibrin(PRF) is a healing biomaterial with a great potential for bone and soft tissue regeneration, without any inflammatory reactions
  Interventions: Procedure: PLATELET RICH FIBRIN in grade II furcation

INTERVENTIONS:
Drug: RhBMP-2 absorbable sponge in grade II furcation — The collagen sponge is impregnated with rhBMP-2 at a concentration of 0.5 μg/ml/1cm3 and were stored at 4°C. This rhBMP-2 impregnated collagen sponge was then dispensed at grade II furcation site
  Other Names: Experimental group
  Arms: RhBMP-2
Procedure: PLATELET RICH FIBRIN in grade II furcation — For preparation of PRF, patient's venous blood is collected into 10ml glass tube or glass-coated plastic tube and centrifuged at 2700 rpm for 12min which leads to two different layers in the test tube, the upper platelet rich fibrin and the lower RBC portion. The formed PRF clot could then be removed from the glass tube and used in grade II furcation
  Other Names: Control group
  Arms: PLATELET RICH FIBRIN

SUMMARY:
The present study evaluated clinically and radiographically the regenerative potential of rhBMP-2 in absorbable sponge and PRF in Grade II furcation.

DETAILED DESCRIPTION:
44 subjects were enrolled in the study. PPD, CAL, plaque index and gingival index were recorded and the evaluation of bone fill was performed after 6 months by using ImageJ® software. After 6 months, the bone fill obtained with rhBMP-2 was higher when compared to PRF. From this trial conducted over a period of 6 months, the unique properties associated with rhBMP-2 in absorbable sponge makes it a potential agent to be used as a graft material for Grade II furcation defects.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy male and female patients of age group 20-55 yrs
* grade II furcation involvement and probing pocket depth of ≥5mm

Exclusion Criteria:

* Medically compromised patients
* subjects who underwent radiotherapy or chemotherapy in the past 12 months
* patients having uncontrolled periodontal disease and
* subjects smoking ≥10 cigarettes per day were excluded

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
BONE FILL | 6 MONTHS
  The evaluation of bone fill was performed after 6 months by using ImageJ® software.

CONTACTS AND LOCATIONS:
Locations (1):
- RV Chandra, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No